CLINICAL TRIAL: NCT01844752
Title: A Multi-Center, Randomized, Evaluator-Blinded, Vehicle-Controlled, Parallel Group, 3-arm Study Comparing the Efficacy, Tolerability and Safety of 2 Concentrations of NVN1000 Gel and Vehicle Gel Twice Daily in the Treatment of Acne Vulgaris.
Brief Title: A Phase 2, 3 Arm Study of NVN1000 Gel and Vehicle Gel in Subjects With Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC201
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NVN1000 1% Gel (Experimental): NVN1000 1% Gel twice daily
  Interventions: Drug: NVN1000 1% Gel
- NVN1000 4% Gel (Experimental): NVN1000 4% Gel twice daily
  Interventions: Drug: NVN1000 4% Gel
- Vehicle Gel (Placebo Comparator): Vehicle Gel twice daily
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: NVN1000 1% Gel — Twice daily NVN1000 1% Gel for 12 weeks
  Other Names: NVN1000
  Arms: NVN1000 1% Gel
Drug: NVN1000 4% Gel — Twice daily NVN1000 4% Gel for 12 weeks
  Other Names: NVN1000
  Arms: NVN1000 4% Gel
Drug: Vehicle Gel — Twice daily Vehicle Gel for 12 weeks
  Other Names: Comparator Gel
  Arms: Vehicle Gel

SUMMARY:
This is a 12 week clinical trial in subjects with acne vulgaris. Subjects will be randomized to NVN1000 1% Gel, NVN1000 4% Gel or Vehicle Gel twice daily. Safety, tolerability and efficacy will be assessed over the course of the study.

DETAILED DESCRIPTION:
This is a multi-center, evaluator and subject blinded, randomized, vehicle-controlled, parallel group, dose-ranging study to be conducted in approximately 150 subjects with acne vulgaris. Subjects who satisfy the entry criteria at the Baseline visit will be randomized to NVN1000 1% Gel, NVN1000 4% Gel or Vehicle Gel in a 1:1:1 ratio. Efficacy assessments will include inflammatory and non-inflammatory lesion counts and investigator global assessments (IGA). Tolerability and safety assessments include cutaneous tolerability evaluation, adverse event collection, physical exams, and laboratory studies. Subjects will return for post-baseline evaluation at Weeks 2, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acne vulgaris and at least 20 but no more than 40 inflammatory lesions, 25-70 non-inflammatory lesions, no more than 2 nodules on the face
* Baseline IGA score of mild, moderate or severe
* Women of child-bearing potential must agree to use an effective method of birth control during the study and for 30 days after their final study visit

Exclusion Criteria:

* Any dermatologic condition or other medical problem that could interfere with clinical evaluation or requires the use of topical or systemic therapy that make evaluations and lesion count inconclusive
* Female subjects who are pregnant, nursing, or considering becoming pregnant
* Methemoglobin > 2% at baseline
* Clinically significant anemia at baseline
* Use of topical or systemic medications to treat acne
* Use of medications that make acne worse, associated with methemoglobinemia, or nitric oxide donors

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The absolute change from baseline in non-inflammatory lesion counts at Week 12 | 12 weeks
  The absolute change from baseline in non-inflammatory lesion counts at Week 12

SECONDARY OUTCOMES:
The absolute change from baseline in inflammatory lesion counts at Week 12 | 12 weeks
  The absolute change from baseline in inflammatory lesion counts at Week 12
Success on the Investigator Global Assessment (IGA) at Week 12 | 12 week
  Analysis of the dichotomized IGA scores (success vs failure) at Week 12. "Success" is defined as a score of "clear" or "almost clear" and a 2 point improvement in the IGA score from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Study Director — Novan, Inc.
Locations (3):
- Instituto Dermatologico & Cirugia de Piel, Santo Domingo, Dominican Republic
- Hospital Y Clinica Bendana, San Pedro Sula, Honduras
- Hosptal Punta Pacifica, Panama City, Panama

REFERENCES:
- [Derived] Baldwin H, Blanco D, McKeever C, Paz N, Vasquez YN, Quiring J, Enloe C, De Leon E, Stasko N. Results of a Phase 2 Efficacy and Safety Study with SB204, an Investigational Topical Nitric Oxide-releasing Drug for the Treatment of Acne Vulgaris. J Clin Aesthet Dermatol. 2016 Aug;9(8):12-8. Epub 2016 Aug 1. PMID 27672413